CLINICAL TRIAL: NCT04099238
Title: Burden of Ischemic Stroke and Adherence to Oral Anticoagulants in Atrial Fibrillation in the UK Primary Care
Brief Title: Burden of Ischemic Stroke and Intake of Oral Anticoagulants in Patients With Atrial Fibrillation in the UK Primary Care
Acronym: BEST-AF
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21094
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation
Keywords: Ischemic stroke; Non-valvular atrial fibrillation (NVAF); Oral anticoagulants (OAC); Vitamin K antagonists (NKA); Non-vitamin K antagonist oral anticoagulants (NOAC); Discontinuation
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke | interventions — Anticoagulants; Warfarin; Acenocoumarol; Phenindione; apixaban; Dabigatran; edoxaban; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with ischemic stroke: Adult subjects from the UK THIN database who were hospitalized for ischemic stroke between 01-Jul-2016 to 30-Jun-2018
  Interventions: Drug: Oral anticoagulant
- NVAF patients with ischemic stroke: Adult subjects from the UK THIN database who were hospitalized for ischemic stroke between 01-Jul-2016 to 30-Jun-2018 and had a diagnosis of NVAF prior to ischemic stroke (Subgroup)
  Interventions: Drug: Oral anticoagulant

INTERVENTIONS:
Drug: Oral anticoagulant — Oral anticoagulants may comprise vitamin K antagonists (VKA) and non-vitamin K antagonist oral antagonists (NOAC).
  Other Names: Warfarin, acenocoumarol, phenindione, apixaban, dabigatran, edoxaban, rivaroxaban

SUMMARY:
This study will characterize patients with ischemic stroke, a condition which occurs when a vessel supplying blood to the brain is obstructed, and a subpopulation of patients with irregular and often rapid heart rate (atrial fibrillation) in a UK general population using The Health Improvement Network (THIN) database.

The main aim of the study is to estimate in how many patients atrial fibrillation was diagnosed at the moment of stroke and to describe whether these patients received OAC at the time of the stroke. In addition, researchers want to learn about the relative risk of ischemic stroke when such patients did not continue OAC treatment.

DETAILED DESCRIPTION:
The primary objectives of the study are to determine the incidence of ischemic stroke in patients registered in the British primary care THIN database and to investigate the OAC exposure, OAC treatment patterns and the relative risk of having an ischemic stroke in relation to OAC treatment for a subgroup of patients, who were diagnosed with non-valvular atrial fibrillation (NVAF) prior to ischemic stroke.

Secondary objectives are to determine the number of patients having NVAF diagnosed at the time of ischemic stroke and within 1 and 12 months after ischemic stroke; to describe cardiovascular risk factors for ischemic stroke and pharmacological treatments before and 12 months after ischemic stroke, and to estimate the case-fatality at 1 and 12 months after the occurrence of ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Occurrence of an ischemic stroke that lead to hospitalization between 01-Jul-2016 to 30-Jun-2018 and concerned adults registered in the THIN database
* Subgroup: Patients with diagnosed NVAF prior or at the time of ischemic stroke

Exclusion Criteria:

* None

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults from UK with electronic medical records in The Health Improvement Network (THIN) database
Sampling Method: Non-Probability Sample
Enrollment: 3739 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Number of subjects with ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2018
Incidence of ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2018
Number of NVAF patients with OAC prescription prior to ischemic stroke | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Duration of OAC treatment before OAC discontinuation for NVAF patients | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Time period from OAC discontinuation to ischemic stroke for NVAF patients | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Relative risk of NVAF patients for ischemic stroke after OAC discontinuation | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Relative risk of NVAF patients for ischemic stroke by time since OAC discontinuation | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Relative risk of NVAF patients for ischemic stroke by OAC treatment duration before OAC discontinuation | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Relative risk of NVAF patients for ischemic stroke after VKA discontinuation | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Relative risk of NVAF patients for ischemic stroke by time since VKA discontinuation | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Relative risk of NVAF patients for ischemic stroke by VKA treatment duration before VKA discontinuation | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Relative risk of NVAF patients for ischemic stroke after NOAC discontinuation | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Relative risk of NVAF patients for ischemic stroke by time since NOAC discontinuation | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only
Relative risk of NVAF patients for ischemic stroke by NOAC treatment duration before NOAC discontinuation | Retrospective analysis of data from 01-Jul-1996 to 30-Jun-2018
  For NVAF subgroup only

SECONDARY OUTCOMES:
Number of subjects with first diagnosis of NVAF at time of ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2018
Number of subjects with first diagnosis of NVAF within 1 month after ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jul-2018
Number of subjects with first diagnosis of NVAF within 12 months after ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019
Prevalence of cardiovascular co-morbidities one year before ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019
Prevalence of cardiovascular co-morbidities 12 months after ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019
Descriptive analysis of pharmacological treatments of patients with known NVAF diagnosis within 12 months before ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019
Descriptive analysis of pharmacological treatments of patients with known NVAF diagnosis within 12 months after ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019
Descriptive analysis of pharmacological treatments of patients without known NVAF diagnosis within 12 months before ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019
Descriptive analysis of pharmacological treatments of patients without known NVAF diagnosis within 12 months after ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019
Case-fatality of patients with known NVAF diagnosis at 1 month after ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019
Case-fatality for patients with known NVAF diagnosis at 12 months after ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019
Case-fatality of patients with unknown NVAF diagnosis at 1 month after ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019
Case-fatality of patients with unknown NVAF diagnosis at 12 months after ischemic stroke | Retrospective analysis of data from 01-Jul-2016 to 30-Jun-2019

CONTACTS AND LOCATIONS:
Locations (1):
- Many facilities, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/